CLINICAL TRIAL: NCT04457830
Title: A Phase 2, Open-label, Single-arm, Multicenter Study of the Efficacy and Safety of F520 in Relapsed/Refractory Peripheral T Cell Lymphoma (PTCL).
Brief Title: The Efficacy and Safety of F520 in Patients With Relapsed/Refractory Peripheral T Cell Lymphoma (PTCL).
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP-F520-002
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-07

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Intervention Model Description: F520
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: F520

INTERVENTIONS:
Drug: F520 — 3mg/kg every 3 weeks

SUMMARY:
It is a multi-center, prospective, open-label, two-stage optimized design, single-arm, phase II clinical study to evaluate the efficacy and safety of F520 for the treatment of relapsed and refractory peripheral T cell lymphoma (PTCL), and to evaluate the immunogenicity of F520.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, male or female;
2. Histologically confirmed relapsed or refractory PTCL patients who had received systemic treatment at least once but had failed to; Relapsed / refractory is defined as follows:

   Relapsed: patients who have new lesions at the primary site or other sites after reaching CR in the previous treatment; Refractory: patients who fail to reach PR in 2 cycles or CR in 4 cycles after first-line or above systemic treatment; if the best effect or end cause is PD, the number of cycles is not required;
3. ECOG score of 0-2;
4. Life expectancy≥3 months;
5. Agree to provide archived tumor tissue samples or fresh tissue samples, including enough samples to complete PD-L1 test;
6. Computed tomography (ct) scans should show the presence of at least one of two vertical orientations; The tumor lesions that could be measured were defined, with the longest diameter of intranode lesion > 1.5cm, the shortest diameter of intranode lesion > 1.0cm and the longest diameter of extranode lesion > 1.0cm;
7. The functions of important organs meet the following requirements (drugs with any blood component and cell growth factor are not allowed to be used within 14 days before the first administration):

   routine blood tests: hemoglobin ≥ 90 g/L, neutrophil ≥ 1.5 ×109/L, platelet ≥ 75×109/L; Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN); If there is liver metastasis, TBIL ≤ 3 × ULN, ALT and AST ≤ 5 × ULN; Serum creatinine ≤ 1.5×ULN; Thyroid function indicators: thyroid-stimulating hormone (TSH) are within the normal range or thyroid-stimulating hormone (TSH) are not within the normal range and free thyroxine (FT3/FT4) are within the normal range;
8. Sign the written informed consent, and be able to follow the visit and related procedures specified in the protocol.

Exclusion Criteria:

1. Diagnosed as vascular immunoblastic t-cell lymphoma (AITL) or adult t-cell lymphoma/leukemia(ATLL);
2. Patients with active central nervous system (CNS) infiltration, including invasion of brain parenchyma, meninges or compression of spinal cord;
3. Diagnosed as cutaneous extranodal nasal type T-cell lymphoma;
4. Immunohistochemistry confirmed PD-1 positive;
5. Patients with complicated diseases, including autoimmune disease, type I diabetes, hypothyroidism requiring hormone replacement (except Hashimoto's thyroiditis) and severe mental disease;
6. The patients received systemic corticosteroids (prednisone > 10 mg/day or equivalent dose) within 2 weeks before the first administration or patients who need systemic corticosteroids therapy during the study;
7. The patients received radiotherapy, chemotherapy, hormone therapy, surgery, targeted therapy or systemic treatment of antibody drugs within 4 weeks before the first administration; the patients used monoclonal antibody coupled radionuclide or cytotoxin therapy within 10 weeks before the first administration; the toxicity of the previous anti-tumor treatment did not recover to ≤ level 1 (except hair loss);
8. Uncontrolled hypertension (systolic blood pressure > 180mmHg and/or diastolic blood pressure > 100mmHg);
9. Previous history of organ transplantation or allogeneic hematopoietic stem cell transplantation;
10. The patients who had autologous hematopoietic stem cell transplantation within 3 months before the first administration;
11. Patients receiving any attenuated vaccine within 4 weeks before the first administration or during the study;
12. Patients who are allergic to macromolecular protein or anti-PD-1 antibody;
13. Patients who with previous or concurrent malignancies (except skin basal cell carcinoma and cervical carcinoma in situ, which have been cured for more than 3 years);
14. Had uncontrollable or serious cardiovascular diseases, the heart of New YorkNYHA standard grade 3-4 history of chronic heart failure, unstable angina, myocardial infarction and other cardiovascular diseases within 6 months before the first administration;
15. HIV positive patients, or active hepatitis (hepatitis B: hepatitis B five items and HBV-DNA, transaminase, etc., hepatitis C: HCV antibody and HCV RNA);
16. Patients who had been previously treated with any other investigational drugs/devices within 4 weeks before the first administration;
17. Patients with drug abuse history or alcohol addiction history within 6 months before the first administration;
18. Patients who were previously treated with anti PD-1 antibody, anti PD-L1 antibody, anti PD-L2 antibody, anti-137 or anti CTLA-4 antibody (or any other antibodies acting on T cell co-stimulation or checkpoint pathway);
19. Patients with current or previous interstitial lung diseases (except for interstitial lung disease caused by radiotherapy and chemotherapy and currently without symptoms);
20. Active infections requiring systemic treatment;
21. Patients with active pulmonary tuberculosis;
22. pregnant or lactating women, female patients with pregnancy plan or male patients with such plan from the study period to 6 months after the last medication, who are unwilling to use an effective contraceptive measure (such as IUD or condom) approved by medicine during the trial period;
23. Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Approximately 24 months
  To evaluate the efficacy of F520 as defined by objective response rate (evaluated by IRC) in patients with relapsed or refractory PTCL.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 24 months
  To evaluate the efficacy of F520 as defined by objective response rate (evaluated by investigator) in patients with relapsed or refractory PTCL.
Completed response rate (CRR) | Approximately 24 months
  To evaluate the efficacy of F520 as defined by completed response rate (evaluated by investigator/IRC) in patients with relapsed or refractory PTCL.
Duration of response (DOR) | Approximately 24 months
  To evaluate the duration of response (DOR) of F520 in patients with relapsed or refractory PTCL.
Overall survival (OS) | Approximately 24 months
  To evaluate the duration from the first administration to death because of any reason in patients with relapsed or refractory PTCL.
Progression-free survival (PFS) | Approximately 24 months
  To evaluate the efficacy of F520 as defined by progression-free survival, in patients with relapsed or refractory PTCL.
Disease control rate (DCR) | Approximately 24 months
  To evaluate the efficacy of F520 as defined by disease control rate, in patients with relapsed or refractory PTCL.
Time to response (TTR) | Approximately 24 months
  To evaluate the efficacy of F520 as defined by time to response in patients with relapsed or refractory PTCL.